CLINICAL TRIAL: NCT00275132
Title: A Randomised, Placebo-Controlled Trial of Erlotinib in Patients With Advanced NSCLC Unsuitable for Chemotherapy
Brief Title: Erlotinib in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Acronym: TOPICAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000457755; LLCG-TOPICAL; EU-20313; ISRCTN (Registry Identifier: 77383050); Cancer Research UK (CTAAC) (Other Grant/Funding Number: C1438/A4147); Roche AG Pharma (Other Grant/Funding Number: MO17591); UCL Trial Sponsor reference (Other: UCL/05/173); EudraCT number (Other: 2004-000729-31)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib (Experimental): Tarceva (OSI-774, erlotinib) PO 150mg daily
  Interventions: Drug: erlotinib hydrochloride
- Matched placebo (Placebo Comparator): Matched placebo PO daily
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: erlotinib hydrochloride — Tarceva (OSI-774, erlotinib) PO 150 mg daily
  Other Names: OSI-774; Tarceva
  Arms: Erlotinib
Drug: Matched placebo — Matched placebo PO daily
  Arms: Matched placebo

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether erlotinib is more effective than a placebo in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying erlotinib to see how well it works compared to a placebo in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare survival of patients with stage IIIB or IV non-small cell lung cancer that is not suitable for first-line chemotherapy treated with erlotinib vs placebo.

Secondary

* Compare progression-free survival and response rate.
* Compare toxicity.
* Compare the quality of life.
* Compare cost-effectiveness.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral erlotinib once daily for up to 24 months.
* Arm II: Patients receive oral placebo once daily for up to 24 months. Quality of life is assessed periodically.

After completion of study treatment, patients are followed periodically for survival.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 664 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Advanced disease (stage IIIB or IV)
  * Diagnosis within 62 days prior to randomization
* Not suitable for first-line chemotherapy, as defined by the following criteria*:

  * ECOG performance status 2-3
  * ECOG performance status 0-1 AND creatinine clearance < 60 mL/min
* NOTE: *These criteria do not imply that all such patients are unsuitable for chemotherapy; patients are considered unsuitable on a case by case basis
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Estimated life expectancy of at least 8 weeks
* Able to take oral medication
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe uncontrolled infection
* No unstable angina
* No myocardial infarction within the past month
* No uncontrolled inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
* No acute renal failure
* Bilirubin < 2 times upper limit of normal (ULN)
* Transaminases < 2 times ULN (5 times ULN if liver metastases are present)
* Creatinine < 5 times ULN
* No evidence of other significant laboratory finding or uncontrolled medical illness that would interfere with study treatment or results comparison or render the patient at high risk from treatment complications
* No other prior or current malignant disease likely to interfere with study treatment or comparisons

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior biological anticancer therapy (e.g., gefitinib, thalidomide, or cetuximab)
* No prior palliative radiotherapy

  * Prior palliative radiotherapy to bone metastases allowed within the past 2 weeks
* No concurrent cyclooxygenase-2 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | between date of randomisation and date of death from any cause

SECONDARY OUTCOMES:
Progression free survival | from the date of randomisation to the date of first clinical evidence of progressive disease, or death.
Adverse events/Toxicity | during and for 28 days following Tarceva/placebo treatment
Quality of life | between randomisation and 8 weeks.
  QL will be measured using the patient-completed EORTC-QLQ C30 and lung cancer module (LC 14). The primary QL outcome measures will be changes in overall QL and the five most commonly reported lung cancer symptoms (fatigue, breathlessness, cough, emotional functioning and pain).
Cost-effectiveness | from date of randomisation to death
  Effectiveness will be estimated in terms of quality-adjusted life years. Mean survival will be calculated on the basis of observed mortality (i.e. a within-trial estimate) and by extrapolating the survival curves if some patients remain alive at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Siow M Lee, MD, PhD, FRCP, Study Chair — University College London Hospitals
Locations (1):
- London Lung Cancer Group, London, England, United Kingdom